CLINICAL TRIAL: NCT01413230
Title: Evaluation of Immunologic Response After Vitamin D Supplementation in Patients With Systemic Lupus Erythematosus
Brief Title: Vitamin D Supplementation in Systemic Lupus Erythematosus
Acronym: VITALUP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: Record AP
Record Dates: First submitted 2011-06-24; First posted 2011-08-10 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-06

CONDITIONS: Vitamin D Deficiency
Keywords: Systemic lupus erythematosus; vitamin D supplementation; regulatory T cells; Th17 cells
MeSH Terms: conditions — Vitamin D Deficiency; Lupus Erythematosus, Systemic | interventions — Cholecalciferol

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood with RNA
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: cholecalciferol — 100 000 UI of cholecalciferol per week during 4 then 100 000 UI of cholecalciferol per month for 6 months
  Other Names: 100 000 UI of cholecalciferol per week during 4; then 100 000 UI of cholecalciferol per month for 6 months

SUMMARY:
Systemic Lupus Erythematosus (SLE) is a systemic autoimmune disorder. It mainly involves the skin, the joints, the nervous system and the kidney and may be life threatening.

SLE is associated with production of autoantibodies and perturbations in regulatory T cells and T helper lymphocytes producing interleukin (IL)-17 (Th17 cells).

Treatments include corticosteroids, hydroxychloroquine and immunosuppressive agents.

Immunomodulatory effects of vitamin D supplementation in VITRO was recently described, notably the expansion of Treg able to suppress inflammatory responses mediated by CD4+ and CD8+ T cells and the decrease of Th17 cells.

DETAILED DESCRIPTION:
Systemic Lupus Erythematosus (SLE) is a systemic autoimmune disorder. It mainly involves the skin, the joints, the nervous system and the kidney and may be life threatening.

SLE is associated with production of autoantibodies and perturbations in regulatory T cells and T helper lymphocytes producing interleukin (IL)-17 (Th17 cells).

Treatments include corticosteroids, hydroxychloroquine and immunosuppressive agents.

Immunomodulatory effects of vitamin D supplementation in VITRO was recently described, notably the expansion of Treg able to suppress inflammatory responses mediated by CD4+ and CD8+ T cells and the decrease of Th17 cells.

Objective : To evaluate the cellular immune response after vitamin D supplementation in patients with SLE.

Methods : This is an open prospective trial. SLE patients with hypovitaminosis D (< 30 ng/mL) receive vitamin D supplementation. 100 000 UI of cholecalciferol per week for 4 weeks then 100 000 UI of cholecalciferol per month for 6 months will be administered. All patients are followed after the beginning of vitamin D supplementation at month 2 and month 6.

End points :

1. Clinical and biological tolerance: Absence of hypercalcemia or lithiasis during and after vitamin D supplementation.
2. Immunologic follow-up of T cells and B cells homeostasis (including Treg and Th17) and gene expression profile in PBMCs using TRANSCRIPTOMIC analysis, before, during and after vitamin D supplementation.
3. Clinical efficacy: follow-up of clinical manifestations of SLE and disease activity score (SLEDAI) during and after vitamin D supplementation.

Schedule : Duration of patients' inclusion period is estimated 3

ELIGIBILITY:
Inclusion Criteria:

* Systemic lupus erythematosus
* Age > 18 years
* Serum vitamin D levels [25(OH)D] < 30 ng/mL
* Low to moderate active disease without modification of associated treatments

Exclusion Criteria:

* Pregnancy
* Serum 25(OH)D levels > 30 ng/mL
* Flare requiring modification of treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with SLE
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Immunologic follow-up of T cells and B cells homeostasis (including regulatory T cells and Th17 cells) and gene expression profile of PBMCs using TRANSCRIPTOMIC analysis, before, during and after vitamin D supplementation | 6 months
  Immunologic follow-up of T cells and B cells homeostasis (including regulatory T cells and Th17 cells) and gene expression profile of PBMCs using TRANSCRIPTOMIC analysis, before, during and after vitamin D supplementation

SECONDARY OUTCOMES:
Clinical tolerance: Absence of Hypercalcemia and lithiasis during and after vitamin D supplementation | 6 months
  Clinical tolerance: Absence of Hypercalcemia and lithiasis during and after vitamin D supplementation
Clinical efficacy: follow-up of clinical manifestations of SLE and disease activity score (SLEDAI) | 6 months
  Clinical efficacy: follow-up of clinical manifestations of SLE and disease activity score (SLEDAI)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Costedoat-Chalumeau, PUPH, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (3):
- France (3):
  - Chu Pitie Salpetriere, Paris
  - Hopital la Pitie Salpétrière, Paris
  - Nathalie Costedoat-Chalumeau, Paris